CLINICAL TRIAL: NCT00297362
Title: Open Observational Study of Galantamine Hydrobromide Administration for the Treatment of Patients With Mild to Moderate Dementia of the Alzheimer Type
Brief Title: A Study of the Safety and Effectiveness of Galantamine Hydrobromide in Patients With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Responsible Party: Medical Affairs Director, Janssen Cilag Pharmaceutica S.A.C.I., Greece
Other Study IDs: CR003559; 57504DEM4001 (Other: Janssen Cilag Pharmaceutica S.A.C.I., Greece)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Dementia; Brain Disease; Memory Loss; Caregiver; Galantamine hydrobromide; Nervous System Diseases; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Memory Disorders; Nervous System Diseases; Mental Disorders | interventions — Galantamine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Galantamine hydrobromide
  Interventions: Drug: Galantamine hydrobromide

INTERVENTIONS:
Drug: Galantamine hydrobromide — 247 patients with diagnosed mild to moderate Alzheimer disease.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of galantamine hydrobromide in patients with Alzheimer's disease who have not received or have not responded to treatment with medication similar to galantamine hydrobromide.

DETAILED DESCRIPTION:
Galantamine hydrobromide is a medication that is approved for the treatment of symptoms of Alzheimer's disease. In accordance with international guidelines, studies are conducted after a drug is marketed to continue to evaluate and expand the knowledge regarding its safety. This is a multi-center, open-label (all people involved know the identity of the intervention), observational study (individuals are observed or certain outcomes are measured - no attempt is made to affect the outcome) to collect information regarding the safety and effectiveness of galantamine hydrobromide in patients with Alzheimer's disease. Patients who have been prescribed galantamine hydrobromide as initial treatment with this type of medication for their Alzheimer's disease or who have failed previous treatment with similar medication of this type for their Alzheimer's disease will receive galantamine hydrobromide for 6 months. The individual physicians responsible for the treatment of Alzheimer's disease will administer galantamine hydrobromide at doses appropriate for each patient and will continue to oversee their care. No medication will be supplied by the sponsor of this study. Safety evaluations (incidence of adverse events, physical exams, vital signs and laboratory tests) will be performed throughout the study. Effectiveness will be determined using standard tests and rating scales to assess mental status, functioning, thinking, behavior, judgment and language (Neuropsychiatric Inventory, [NPI], Mini Mental Status Exam [MMSE] and Clinical Global Impression-Caregiver [CGI-Caregiver]). Assessments will be conducted monthly for the first 3 months and at the end of 6 months of treatment. Galantamine hydrobromide treatment should be discontinued if there is no further indication of effectiveness. At the end of the study, the treating physician may continue treatment with galantamine hydrobromide in responding patients as appropriate. The study hypothesis is that galantamine hydrobromide will be effective in treating the symptoms associated with Alzheimer's disease and is safe and well-tolerated. Observational study -No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients with a score of 10-26 on the Mini Mental Status Exam
* Patients who have not yet received treatment for their Alzheimer's disease with a medication similar to galantamine or patients who have been treated with as medication similar to galantamine hydrobromide and who have discontinued that medication due to lack of effectiveness or poor tolerability (adverse events)

Exclusion Criteria:

* Patients with severely decreased liver or kidney function
* Patients with a digestive system or urinary blockage who are recovering from digestive system or urinary bladder surgery
* Patients with clinically significant unstable or uncontrolled hormonal or mental disease
* Patients who are unable to take the medication either alone or with help from another person who is available during the entire study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 247 patients with diagnosed with mild to moderate Alzheimer's disease with a score of 10-26 on the Mini Mental Status Exam. Patients switching from an acetylcholinesterase inhibitor treatment due to lack of efficacy or poor tolerability.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2004-06; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Mini-Mental State Examination (MMSE) scale scores | Baseline to 6 months
  The MMSE is a brief 30-point questionnaire test that is used to screen for cognitive impairment. A score greater than or equal to 25 points is effectively normal (intact). Below this, scores can indicate severe (≤9 points), moderate (10-20 points) or mild (21-24 points) cognitive impairment.
Changes from baseline in Disability Assessment for Dementia (DAD) scale scores | Baseline to 6 months
  The 40-item DAD scale assesses functional abilities in activities of daily living in patients with dementia and other cognitive impairments. Higher scores indicate less disability while lower scores denote more difficulties.
Changes from baseline in Neuropsychiatric Inventory (NPI) scale scores | Baseline to 6 months
  The NPI assesses psychopathology in dementia patients. It evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. Both the frequency (from rarely to very often) and the severity (from mild to severe) of each behavior are determined.
Changes from baseline in Clinical Global Impression (CGI) scale scores | Baseline to 6 months
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients".
Changes from baseline in Cornell Scale | Baseline to 6 months
  The Cornell Scale assesses signs and symptoms of major depression in patients with dementia. Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 as a rule are associated with absence of significant depressive symptoms.

SECONDARY OUTCOMES:
Number of patients with Adverse Events as Measure of Safety and Tolerability | 6 months
Number of patients whose vital signs fell outside the normal ranges | 6 months
Number of patients whose laboratory test results fell outside the normal ranges | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.

REFERENCES:
- See also: Open Observational Study of Galantamine Hydrobromide Administration for the Treatment of Patients with Mild to Moderate Dementia of the Alzheimer Type — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=256&filename=CR003559_CSR.pdf